CLINICAL TRIAL: NCT01153399
Title: An NIS Registry for the Epidemiological and Scientific Evaluation of EGFR Mutation Status in Patients With Newly Diagnosed Locally Advanced or Metastatic NSCLC (Stage IIIB/IV Non-small Cell Lung Cancer)-REASON STUDY.
Brief Title: A Non-interventional Study (NIS) Registry for the Epidemiological and Scientific Evaluation of Epidermal Growth Factor Receptor (EGFR) Mutation Status in Patients With Newly Diagnosed Locally Advanced or Metastatic Non Small Cell Lung Cancer (NSCLC) (Stage IIIB/IV Non-small Cell Lung Cancer).
Acronym: REASON
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-OGR-DUM-2010/1
Record Dates: First submitted 2010-06-25; First posted 2010-06-30 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Non Small Cell Lung Cancer; EGFR mutations
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with Non Small Cell Lung Cancer, visiting hospital oncology clinics

SUMMARY:
The primary objective of the study is to collect epidemiological data on EGFR mutation status [M+(mutation positive), M-(mutation negative)] in a population of predominantly Caucasian ethnicity, and to correlate EGFR mutation status with clinico-pathological characteristics (e.g. smoking status, sex, histology, etc). In particular, the study will aim to determine the frequency of EGFR M+ lung cancers in patients with clinico-pathological characteristics that are not commonly associated with EGFR mutation positivity (i.e., smokers, men, and non-adenocarcinoma).

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent.
2. Female or male aged 18 years or above.
3. Histologically confirmed locally advanced or metastatic NSCLC (stage IIIB/IV).
4. Patients receiving 1st-line treatment for IIIB/IV NSCLC.
5. Patients with known EGFR mutation status (i.e. patients must be either EGFR M+, EGFR M- or EGFR Mx).
6. Tumour not amenable to curative surgery or radiotherapy.

Exclusion Criteria:

1. Mixed histology of small cell and non-small cell lung cancer.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Non Small Cell Lung Cancer
Sampling Method: Probability Sample
Enrollment: 589 (Actual)
Dates: Start 2010-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Epidemiological data on EGFR mutation status (M+, M-) in a population of predominantly Caucasian ethnicity | Up to 2,5 years
Clinico-pathological characteristics according to mutation status | Up to 2,5 years

SECONDARY OUTCOMES:
Pharmacoeconomic data (resource use) associated with the diagnosis and treatment of EGFR M+ patients | Up to 3,5 years
Real-life data on 1st-line treatment decisions in EGFR M+ and M-/Mx(mutation status not evaluable) patients | Up to 2,5 years
Clinical outcome data under real life clinical practice in all EGFR M+ patients up to disease progression (PFS, OS, DCR) | Up to 3,5 years

CONTACTS AND LOCATIONS:
Overall Officials: Panagiotis Pontikis, Study Director — AstraZeneca
Locations (9):
- Greece (9):
  - Research Site, Athens, Athens
  - Research Site, Crete, Crete
  - Research Site, Ioannina, Ioannina
  - Research Site, Kavala, Kavala
  - Research Site, Larissa, Larisa
  - Research Site, Pátrai, Patra
  - Research Site, Ptolemaida, Ptolemaida
  - Research Site, Thessaloniki, Thessaloniki
  - Research Site, Volos, Volos

REFERENCES:
- See also: CSR_Synopsis_NIS-OGR-DUM-2010_1.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=998&filename=CSR_Synopsis_NIS-OGR-DUM-2010_1_version_1_0_abstract.pdf